CLINICAL TRIAL: NCT03180372
Title: Safety and Efficacy of Hybrid Fractional Laser diVa Treatment for Symptoms of Urinary Incontinence
Brief Title: Hybrid Fractional Laser Treatment for Symptoms of Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIVACIP001
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence; Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hybrid Fractional Laser (Experimental): Hybrid fractional 2940 nm and 1470 nm laser treatment
  Interventions: Device: Hybrid Fractional Laser

INTERVENTIONS:
Device: Hybrid Fractional Laser — Consecutive and coincident fractional 2940 nm and 1470 nm lasers
  Other Names: diVa

SUMMARY:
This multi-center clinical trial will evaluate the safety and long-term efficacy of hybrid fractional 2940 nm and 1470 lasers for improvement of symptoms of urinary incontinence.

DETAILED DESCRIPTION:
Both 2940 nm Er:YAG (Erbium-doped yttrium aluminium garnet) and 1470 nm diode lasers are cleared by the Food and Drug Administration (FDA) for ablation, vaporization, coagulation of soft tissue and for skin resurfacing. Fractional delivery of laser is a well-established method that stimulates tissue remodeling in the dermis while leaving the surrounding tissue intact in order to decrease healing time. The layers of skin and vaginal mucosal tissue exhibit similarities that suggest the clinical results seen with skin resurfacing may be translated to the vaginal tissue. Improved vaginal tissue tone and increased collagen formation in the lamina propria beneath the urethra may lead to improved urinary control. This multi-centered, 18-month prospective clinical trial will determine the safety and long-term effectiveness of hybrid fractional 2940 nm and 1470 nm lasers (Hybrid Fractional Laser) as an alternative non-surgical, non-hormonal treatment for improvement of symptoms of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy biological female aged between 30 to 75 years
2. Is experiencing at least one or a combination of the following symptoms of urinary incontinence (UI)

   1. involuntary urine leakage on effort, exertion, sneezing, coughing
   2. sudden intense urge to urinate followed by involuntary loss of urine
3. Has been experiencing symptoms of UI for greater than 3 months
4. Normal urinalysis
5. Has indicated willingness to participate in the study by signing an informed consent form
6. Can read, understand and sign informed consent form
7. Agree to adhere to the treatment and follow-up schedule and post treatment care instructions

Exclusion Criteria:

1. Undiagnosed abnormal genital bleeding
2. Has history of pelvic surgery or other energy-based vaginal therapy within 6 months prior to enrollment
3. Is pregnant or planning to get pregnant within the study period
4. Is currently breastfeeding
5. Has an active sexually transmitted infection (STI)
6. Has equal to or greater than stage III prolapse, according to pelvic organ prolapse quantification system (POP-Q test)
7. Has signs or symptoms of vaginitis/vulvitis
8. Has signs or symptoms of acute urinary tract infection (UTI)
9. Has voiding dysfunction or urinary retention
10. Has predominantly overactive bladder (OAB) as proven by urodynamics
11. Is currently taking medication for treating urinary incontinence
12. Has a known history of neurologic disease
13. Has history of heart failure
14. Any medical conditions that might interfere with wound healing
15. Has history of abnormal wound healing
16. Has participated in any clinical trial involving an investigational drug or procedure within past 30 days
17. The investigator feels that for any reason the subject is not eligible to participate in the study.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Cough Stress Test | 14 months
  A diagnostic test to simulate accidental release of urine when the patient coughs.

SECONDARY OUTCOMES:
Change from baseline in Incontinence Impact Questionnaire (IIQ-7) | 14 months
  A 7-item self-report instrument designed to assess the impact of urinary incontinence on a patient's life.
Change from baseline in Urogenital Distress Inventory (UDI-6) | 14 months
  A 6-item self-report instrument that assesses symptom distress and the impact on daily life of urinary incontinence.
Change from baseline in Female Sexual Function Index (FSFI) | 14 months
  A multidimensional self-report instrument for assessment of female sexual function.
Change from baseline in Histology | 14 months
  Change from baseline in epithelial thickness, collagen, elastin, vascularity, and fibroblast density.
Change from baseline in Urodynamic Testing | 14 months
  Quantitative measures of uroflowmetry, post-void residual (PVR) urine, cystometry, leak-point pressure, pressure flow, urethral pressure profile, and the functional urethral length.
Incidence and severity of treatment-related Adverse Events | 14 months
  Incidence and severity of treatment-related adverse events (i.e. pain, edema, erythema, altered sensation, scarring, and/or potential infection).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Women's Pelvic Health Institute, Los Gatos, California
  - Coyle Institute, Pensacola, Florida
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Woodlands Gynecology & Aesthetics, The Woodlands, Texas
  - The Female Pelvic Medicine Institute of Virginia, North Chesterfield, Virginia

IPD SHARING:
Plan to Share IPD: No